CLINICAL TRIAL: NCT05989243
Title: Improving Socket Fit in Female and Male Veterans With Transtibial and TransfemoralAmputation
Brief Title: Improving Socket Fit in Female and Male Veterans With Transtibial and Transfemoral Amputation
Acronym: SocketFit
Status: Recruiting | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: A3643-R
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Transtibial Amputation; Transfemoral Amputation
Keywords: Biomechanics; Kinematics; Walking; Prostheses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Veterans with a transtibial amputation: 20 Veterans with a transtibial amputation, 10 females and 10 males
  Interventions: Device: Conventional prosthetic socket; Device: Adjustable Quatro socket
- Veterans with a transfemoral amputation: 20 Veterans with a transfemoral amputation, 10 females and 10 males
  Interventions: Device: Conventional prosthetic socket; Device: Adjustable Quatro socket

INTERVENTIONS:
Device: Conventional prosthetic socket — Participants will use their own conventional rigid socket and will be asked to walk on a force-measuring treadmill on level ground at 0.75, 1.0, 1.25, and 1.5 m/s for ~60 sec per speed. They will also be asked to evaluate this socket using a questionnaire.
Device: Adjustable Quatro socket — Participants will use an adjustable Quatro socket and will be asked to walk on a force-measuring treadmill on level ground at 0.75, 1.0, 1.25, and 1.5 m/s for ~60 sec per speed. They will also be asked to evaluate this socket using a questionnaire.

SUMMARY:
The investigators do not yet know how a prosthetic socket with adjustable panels affects the performance of people with a lower limb amputation compared to a conventional prosthetic socket. The primary objective of this study is to compare an adjustable and conventional prosthetic socket and use this information to determine the optimal socket that would improve rehabilitation and function in people with lower limb amputation.

DETAILED DESCRIPTION:
The purpose of the project is to determine the effects of using different prosthetic socket designs with the same suspension and components on the biomechanical asymmetry, residual limb movement within the socket (socket pistoning) and comfort/satisfaction of 20 Veterans with a transtibial amputation and 20 Veterans with a transfemoral amputation, 10 males and 10 females per group.

ELIGIBILITY:
Inclusion Criteria:

* The investigators will enroll up to 40 Veterans

  * 20 with unilateral transtibial amputation
  * 20 with unilateral transfemoral amputation who are at or above a K2 Medicare functional classification level (MFCL) and who are 18-65 years old
* All participants will have no current problems with their prosthesis or residual limb, and be at least 6-months post-amputation
* Participants will be at or above a K2 MFCL, defined as a person who has the ability or potential for ambulation with the ability to traverse low level environmental barriers such as curbs, stairs, or uneven surfaces, typical of the limited community ambulator

Exclusion Criteria:

* Cardiovascular, pulmonary, or neurological disease or disorder or requirement for an assistive device for their unaffected leg (i.e. orthosis, cane)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20 Veterans with unilateral transtibial amputation and 20 Veterans with unilateral transfemoral amputation
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Biomechanical Asymmetry | through study completion, an average of 4 years
  The assessments of ground reaction forces, and joint motion, torque, power, and work will be aggregated into a measure of asymmetry that compares the percentage difference between the affected and unaffected legs of each participant. The investigators will compare asymmetry between groups and sockets.
Prosthetic Evaluation Questionnaire | through study completion, an average of 4 years
  The prosthetic evaluation questionnaire assesses comfort and satisfaction. This questionnaire asks participants to rate their comfort and satisfaction based on a 10-point scale and contains 54 questions organized into 9 domain scales, where each scale can be used to independently measure a domain. The investigators will compare overall and domain-specific scores between groups and sockets.

SECONDARY OUTCOMES:
Socket pistoning | through study completion, an average of 4 years
  Movement of the residual limb within the socket. The investigators will compared socket pistoning between groups and sockets.

CONTACTS AND LOCATIONS:
Overall Officials: Alena Grabowski, PhD BA, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No